CLINICAL TRIAL: NCT00873535
Title: Effect of Varenicline on Reactivity to Smoking and Drinking Cues in Individuals With Concurrent Tobacco Dependence and Alcohol Use
Brief Title: Effect of Varenicline on Reactivity to Smoking and Drinking Cues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Laurie Zawertailo, Clinical Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 114/2008
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Tobacco Dependence; Alcohol Dependence
Keywords: Nicotine; Nicotine dependence; Smoking cessation; Alcohol; Alcohol dependence; Alcohol cessation; Treatment; Smoking; Cigarette; Heavy drinkers; Social drinkers; Co-morbidity of alcohol and nicotine dependence; Nicotine receptor; Nicotinic receptor; Nicotinic acetycholine receptor; Alpha-4-beta-2 nicotinic acetycholine receptor; Cholinergic receptor; Dopamine; Craving; Diary; Cue induced; Pharmacotherapy; Varenicline; Chantix; Champix
MeSH Terms: conditions — Tobacco Use Disorder; Alcoholism; Smoking Cessation; Smoking | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Active Comparator): This group (N=40) will receive Varenicline (0.5mg once daily for days 1-3, 0.5mg twice daily for days 4-7 followed by 1mg twice daily for days 8-14). The group will consist of heavy smokers and heavy drinkers (N=20) and heavy smokers and social drinkers (N=20).
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): This group (N=40) will receive placebo in the same dosing regimen as for Varenicline. The group will consist of heavy smokers and heavy drinkers (N=20) and heavy smokers and social drinkers (N=20).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — This group (N=40) will receive Varenicline (0.5mg once daily for days 1-3, 0.5mg twice daily for days 4-7 followed by 1mg twice daily for days 8-14). The group will consist of heavy smokers and heavy drinkers (N=20) and heavy smokers and social drinkers (N=20).
  Other Names: Chantix; Champix
  Arms: Varenicline
Drug: Placebo — This group (n=40) will receive matching placebo capsules in the identical dosing regimen described for the Varenicline arm. The group will consist of heavy smokers who are heavy drinkers (n=20) and heavy smokers who are social drinkers (n=20).
  Arms: Placebo

SUMMARY:
Alcohol and nicotine dependence are often co-morbid, with 85% of alcoholics also smoking. However, very little research has been conducted into the nature of this co-occurrence. Thus, the main aim of this study is to assess differences in alcohol and tobacco consumption and cue-induced craving in treatment-seeking smokers after two weeks treatment of varenicline.

Hypotheses

1. Two weeks of varenicline treatment will significantly decrease cue-induced tobacco craving compared to placebo (Due to the actions of varenicline on alpha-4-beta-2 receptors and its downstream effect on dopamine release).
2. Varenicline will decrease cue-induced alcohol craving compared to placebo.
3. The impact of Varenicline on cue-induced alcohol craving will be greater in heavy drinkers compared to social drinkers.

DETAILED DESCRIPTION:
The relationship between alcohol and tobacco dependence needs to be addressed as such populations are generally excluded from clinical trials involving smoking cessation pharmacotherapy. Furthermore, the effect of Varenicline(Pfizer Pharmaceuticals)treatment on tobacco cue-induced craving has not been empirically measured, nor has the effect of varenicline on alcohol consumption. In addition to being an effective aid in smoking cessation, preliminary evidence has shown that Varenicline can decrease alcohol consumption in animal models.

Varenicline is a partial agonist of the α4β2 nicotinic acetylcholine receptor. This drug's partial agonist effect allows for the activation of this receptor at a lesser degree than nicotine while simultaneously preventing nicotine binding due to the drugs high affinity (i.e.: antagonist effect) for this receptor subtype.

Varenicline has recently been approved in Canada as an aid for smoking cessation. This study will be a double-blind, placebo-controlled randomized study. It will assess differences in alcohol and tobacco consumption and cue-induced craving in treatment-seeking smokers after two weeks of treatment with either varenicline or placebo.Ultimately This study may help to further understand the association between smoking and drinking alcohol.

This study will consist of two study groups composed of 40 subjects each being randomized to receive either placebo or varenicline (0.5mg once daily for days 1-3, 0.5mg twice daily for days 4-7 followed by 1mg twice daily for days 8-14). One group will be heavy smokers and heavy drinkers while the other will be heavy smokers and social drinkers. Upon entering the study, subjects will undergo baseline cognitive and craving measures for both tobacco and alcohol associated cue presentations prior to randomization to varenicline or placebo. Subjects will be provided a 1-week supply of study medications and directions for use. During this period, subjects will be requested to complete a diary outlining their cigarette and alcohol craving and consumption each day and outline any adverse effects. Upon completion of this 1-week period, subjects will attend the Centre for Addiction and Mental Health (CAMH) where their old pill bottles and daily diaries will be collected and they will be supplied with study medication (1mg varenicline taken twice daily or placebo) and daily diary for an additional week. At this visit, subjects will complete the symptom checklist. At the end of the second week of treatment, subjects will be requested to return to CAMH where craving for tobacco and alcohol and cue-reactivity will be assessed in a similar manner as to study day After study completion, all subjects will be given the option to continue with varenicline in a 12-week treatment plan through the Nicotine Dependence Clinic.

ELIGIBILITY:
Inclusion Criteria: Heavy Smokers/Heavy Drinkers

* Treatment seeking smokers
* Age 18 to 65 years
* Smoke ≥ 10 cigarettes per day
* Fagerstrom Test of Nicotine Dependence score > 3
* Alcohol Use Disorders Identification Test (AUDIT) > 8
* Drink > 25 drinks per week for males or > 20 drinks per week for females
* Able to provide written informed consent

Inclusion Criteria (Heavy Smokers/Social Drinkers):

* Treatment seeking smokers
* Age 18 to 65 years
* Smoke ≥ 10 cigarettes per day
* Fagerstrom Test of Nicotine Dependence score > 3
* Alcohol Use Disorders Identification Test(AUDIT) < 8
* Drink < 14 drinks per week for males or < 9 drinks per week for females
* Able to provide written informed consent

Exclusion Criteria (Heavy Smokers/Heavy Drinkers):

* Any medical condition requiring immediate investigation or treatment
* Beck Depression Inventory score >16
* Insulin-dependent diabetes
* Drink > 70 standard alcoholic drinks per week for males or drink > 52 standard alcoholic drinks per week for females
* Pregnancy or lactation
* Current DSM-IV Axis 1 psychiatric disorder
* Regular use of any therapeutic or recreational psychoactive drug use during the last three months or other substance use disorder, with the exception of tobacco and alcohol.

Exclusion Criteria (Heavy Smokers/Social Drinkers):

* Any medical condition requiring immediate investigation or treatment
* Beck Depression Inventory score >16
* Insulin-dependent diabetes
* Drink > 14 standard alcoholic drinks per week for males or > 9 standard alcoholic drinks per week for females
* Pregnancy or lactation
* Current DSM-IV Axis 1 psychiatric disorder
* Regular use of any therapeutic or recreational psychoactive drug use during the last three months or other substance use disorder, with the exception of tobacco.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2008-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The Questionnaire of Smoking Urges and the Alcohol Craving Questionnaire. (This questionnaire is used following visual cue presentation consisting of smoking, drinking and neutral pictures). | day 1, day 14

CONTACTS AND LOCATIONS:
Overall Officials: Usoa E. Busto, Pharm.D., Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- [Background] Acheson A, Mahler SV, Chi H, de Wit H. Differential effects of nicotine on alcohol consumption in men and women. Psychopharmacology (Berl). 2006 May;186(1):54-63. doi: 10.1007/s00213-006-0338-y. Epub 2006 Mar 25. PMID 16565827
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.net/research